CLINICAL TRIAL: NCT05423457
Title: Effectiveness of Vegan Diet and MyPlate Diet (Taiwanese Version) on Lipoproteins, Novel Markers of Cardiovascular Diseases, and Traditional Cardiometabolic Risk Factors
Brief Title: Diets, Lipoproteins and Inflammation Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB106-92-B
Record Dates: First submitted 2022-05-30; First posted 2022-06-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2019-06

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome; Diet, Healthy; Vegan Diet; Inflammatory Response
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome | interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan diet (Experimental): Participants were provided with and instructed to eat these foods:
  * flaxseed meal,
  * walnuts,
  * pecans,
  * extra-virgin olive oil,
  * Brazil nuts
  * Taiwanese purple laver (also known as "hong-mao-tai" or Bangia atropurpurea, and was selected to test for its vitamin B12 bioavailability).
  Each Participant has three group sessions and three individual nutrition counseling with a dietitian.
  Interventions: Behavioral: Vegan diet
- MyPlate (Taiwanese version) (Active Comparator): Each Participant has three group sessions and three individual nutrition counseling with a dietitian.
  Interventions: Behavioral: Vegan diet

INTERVENTIONS:
Behavioral: Vegan diet — The participants were advised to eat foods in their original type.

SUMMARY:
Systematic inflammation and lipid profiles are two major therapeutic targets for cardiovascular diseases. The effectiveness of vegan diet has been reported (doi: 10.3389/fnut.2022.807810).

Aim:

To compare the effectiveness of a nutritionally balanced vegan diet and a Myplate diet ((Taiwanese version) on systematic inflammation and lipoprotein subclass.

Design: Randomized crossover design

ELIGIBILITY:
Inclusion Criteria:

Patients with dyslipidemia (at least one of the following)

* TG ≥ 150 mg/dL
* TC ≥ 200 mg/dL
* LDL-c≥ 130 mg/dL,
* HDL-c < 45 mg/dL for male or < 55 mg/dL for female or receiving statin treatment

Exclusion Criteria (fulfill one of the following condition):

* chronic kidney disease
* history of coronary artery disease
* ischemic heart disease,
* heart failure,
* stroke,
* cancer of any type

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Novel inflammatory markers for cardiovascular disease and Lipoprotein particles concentration | 12 weeks
  GlycA (umol/L), lipoprotein particles concentration(umol/L)
Lipoprotein particles concentration | 12 weeks
  lipoprotein particles concentration (nmol/L）
lipoprotein particles size | 12 weeks
  lipoprotein particles size (nm)
Trimethylamine-N-oxide | 12 weeks
  TMAO (uM). TMAO is a low molecular weight compound that belongs to the class of amine oxides
Traditional cadiometabolic risk factors 1 | 12 weeks
  TG(mg/dL), LDL-C(mg/dL), HDL-C(mg/dL), Total cholesterol(mg/dL)
Traditional cadiometabolic risk factors 2 | 12 weeks
  HbA1c(%)
Traditional cadiometabolic risk factors 3 | 12 weeks
  HOMA-IR index (Homeostasis Model Assessment-Insulin Resistance index)

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No